CLINICAL TRIAL: NCT00143481
Title: A Multi-Center, Double-Phase, Randomized, Double-Blind, Placebo Controlled (12-Week Double-Blind Followed by 12-Week Open-Label) Study Evaluating the Effect of Tolterodine ER on Urgency Urinary Incontinence (UUI), Urgency, Frequency, Sexual Quality of Life and Sexual Function in Women With Overactive Bladder
Brief Title: Effect of Detrol LA on Overactive Bladder Symptoms, Sexual Quality of Life and Sexual Function in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121002
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: Tolterodine ER 4mg QD

SUMMARY:
The purpose of the study is to assess the impact of treatment with tolterodine ER versus placebo on Urgency Urinary Incontinence in sexually active women with OAB symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatients 18 years or older.
* Overactive bladder symptoms (subject-reported) for greater than or equal to 3 months.
* Currently sexually active with a male partner.

Exclusion Criteria:

* Diagnosed or suspected interstitial cystitis, uninvestigated hematuria, urogenital cancer, and interstitial or external radiation to the pelvis or external genitalia or clinically significant bladder outlet obstruction.
* Symptoms of incontinence being predominately stress urinary incontinence as determined by the investigator.
* Treated with antimuscarinic/ anticholinergic medication, for any reason including OAB, within the last 3 months or are expected to start therapy during the study treatment period.
* Any drug for urgency urinary incontinence (UUI) initiated within the past 3 months prior to Visit 1, with the exception of estrogen (topical or systemic) as long as treatment is not initiated within 4 weeks prior to Visit 1 (screening)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-03; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change in number of episodes of urgency urinary incontinence (UUI) at week 12 compared with baseline.

SECONDARY OUTCOMES:
Change in total number of urgency urinary incontinence (UUI) episodes at weeks 4 and 24 compared with baseline
Change in total number of daytime urgency urinary incontinence (UUI) episodes at week 4, week 12, and week 24 compared with baseline
Change in total number of pads used per 24 hours at weeks 4, 12, and 24 compared with baseline
Reasons for treatment withdrawal
Adverse Events during the 24 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- United States (49):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, West Hartford, Connecticut
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Leesburg, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Weston, Florida
  - Pfizer Investigational Site, Alpharetta, Georgia
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Saginaw, Michigan
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, North Las Vegas, Nevada
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, New Bern, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Gallipolis, Ohio
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Conroe, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Morgantown, West Virginia

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Rogers RG, Bachmann G, Scarpero H, Jumadilova Z, Sun F, Morrow JD, Guan Z, Bavendam T. Effects of tolterodine ER on patient-reported outcomes in sexually active women with overactive bladder and urgency urinary incontinence. Curr Med Res Opin. 2009 Sep;25(9):2159-65. doi: 10.1185/03007990903103279. PMID 19601704
- [Derived] Rogers R, Bachmann G, Jumadilova Z, Sun F, Morrow JD, Guan Z, Bavendam T. Efficacy of tolterodine on overactive bladder symptoms and sexual and emotional quality of life in sexually active women. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Nov;19(11):1551-7. doi: 10.1007/s00192-008-0688-6. Epub 2008 Aug 7. PMID 18685795
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121002&StudyName=Effect+of+Detrol+LA+on+Overactive+Bladder+Symptoms%2C+Sexual+Quality+of+Life+and+Sexual+Function+in+Women